CLINICAL TRIAL: NCT05734118
Title: Indocyanine Green Fluorescence Angiography Mediated Assessment of Gastro-Intestinal Perfusion in Neonates
Brief Title: Safety and Feasibility of Indocyanine Green Fluorescence for Intraoperative Assessment of Intestinal Perfusion in Young Infants and Neonates
Acronym: IMAGINE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: UMC Utrecht (Other); Stryker Endoscopy (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IMAGINE
Record Dates: First submitted 2022-11-27; First posted 2023-02-17 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: NEC; Atresia; Malrotation; Intestinal Perforation
Keywords: Neonate; Infant; ICG; Fluorescence; Image-guided surgery; Pediatric Surgery; Intestinal perfusion; Anastomosis; Safety; Feasibility; Bowel ischemia
MeSH Terms: conditions — Volvulus Of Midgut; Intestinal Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Intraoperative perfusion assessment using ICG-FA (Experimental): Surgical procedure within standard of care. Intraoperatively, the vitality of the bowel will be assessed visually (the conventional method). Afterwards, participants will be administered indocyanine green intravenously.
  Interventions: Device: Perfusion assessment by means of the SPY-PHI camera

INTERVENTIONS:
Device: Perfusion assessment by means of the SPY-PHI camera — Minutes after injection of ICG, the intestinal perfusion can and will be assessed using the SPY-PHI camera by Stryker Endoscopy. The operative plan will not be changed based on the results of the perfusion assessment. Images will be recorded and evaluated postoperatively.

SUMMARY:
The goal of this clinical trial is to test the use of the SPY-PHI device for the purpose of ICG-mediated intestinal perfusion visualization during gastrointestinal surgery in neonates and young infants (<3 months old) undergoing surgery for NEC, atresia, SIP or malrotation. The main question[s] it aims to answer are:

* Is ICG-FA feasible for intraoperative use in neonates and young infants undergoing laparotomy for NEC, atresia, SIP or malrotation?
* Is ICG-FA is safe to use in neonates during surgery?

Participants will undergo surgical care for their diseases within the standard of care. During laparotomy, the pediatric surgeon will assess bowel perfusion in two ways. First, by visual inspection (the conventional method). Second, the intestine will be analyzed with indocyanine green fluorescence angiography (ICG-FA) by means of the hand-held SPY-PHI camera. For this purpose, the patients will be administered ICG intravenously. Afterwards, the intestinal perfusion will be assessed by means of the SPY-PHI device in 5 to 10 minutes.

Specifically, the feasibility and safety for use of ICG-FA in neonates undergoing laparotomy as treatment for necrotizing enterocolitis (NEC), atresia, spontaneous intestinal perforation (SIP) and malrotation will be investigated.

If ICG-FA turns out to be feasible and safe for the population investigated in this study, a follow-up study will be conducted with the aim to explore the potential benefits of this technique on the postoperative outcome and intraoperative decision-making.

DETAILED DESCRIPTION:
This study aims to investigate whether the intraoperative use of indocyanine green fluorescence angiography (ICG-FA) is feasible and safe in neonates. Feasibility is therein defined as practically possible use of ICG-FA, resulting in clear and interpretable results, with the future potential to improve clinical outcome and benefits for the patient.

Specifically, the feasibility and safety for use of ICG-FA in neonates undergoing laparotomy as treatment for necrotizing enterocolitis (NEC), atresia, spontaneous intestinal perforation (SIP) and malrotation will be investigated.

If ICG-FA turns out to be feasible and safe for the population investigated in this study, a follow-up study will be conducted with the aim to explore the potential benefits of this technique on the postoperative outcome and intraoperative decision-making.

The primary endpoint of this study is assessing the feasibility and safety of intraoperative ICG-FA imaging in neonates undergoing laparotomy for NEC, atresia, SIP, or malrotation. The secondary endpoint of this study is postoperative comparison of the images; standard visual inspection (conventional image) with the corresponding fluorescence image.

During laparotomy, first the pediatric surgeon performs the visual inspection of the predetermined areas (mid jejunum, ileum, ascending colon and sigmoid) as well as regions of interest such as ischemic lesions in NEC and malrotation with volvulus. In case of intestinal necrosis, both edges of the parts that will be resected must be marked with a suture. Second, the intestine will be analyzed using ICG-FA. This analysis will cover the predetermined areas as well as regions of interest.

To this end, the ICG should be injected intravenously by the one member of the anesthetic team. This will only be done if the operating team, consisting of both the consultant surgeon and consultant pediatric anesthesiologist, consider it safe to do so. Utilizing the mobile unit with computer and camera head, the fluorescence angiography system can measure tissue perfusion. Before the start of the procedure in which the SPY-PHY camera will be used intraoperatively, the camera will be covered with sterile drapes. The pediatric surgeon will first make conventional video images with the camera of the predetermined areas and the region of interest and second, the surgeon will make images of the ICG-FA with the camera, which both will be recorded to be analyzed later.

The ICG-FA images do not alter the decision on what type of surgical procedure will be performed and/or how much length of bowel will be resected. In case of a difficult decision, a second pediatric surgeon will be consulted, which is routine clinical practice in both centers anyway.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained by both patient's parents or legal guardians (as applicable);
* Patient is a neonate (< 1 month of age) or young infant (<3 months of age);
* Patient is suffering from necrotizing enterocolitis, atresia, malrotation or spontaneous intestinal perforation;
* Patient requires laparotomy for management of the disease.

Exclusion Criteria:

* Patient is suffering from clinically significant (treatment necessary) hyperbilirubinemia;
* Patient is suffering from thyroid or liver disease;
* Patient is allergic to the active substance indocyanine green or sodium iodide or iodine;
* Patient has abdominal wall defects;
* Patient can be treated non-surgically;
* During the preoperative multidisciplinary meeting with the team, including the pediatric anesthetist, patient is deemed not stable enough hemodynamically to perform the ICG-FU measurements
* Patient is assessed unstable by operating team intraoperatively.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility of ICG-FA for intraoperative assessment of intestinal perfusion | 10 minutes intraoperatively (recording)
  a. Possibility for the researchers to assess intestinal perfusion based on the intraoperative ICG-FA images (clarity: yes/no);
Feasibility of ICG-FA for intraoperative assessment of intestinal perfusion | 10 minutes intraoperatively (recording)
  b. Possibility for the researchers to point out a specific location for resection of the bowel based on visualization of perfusion in the ICG-FA images (interpretability: yes/no);
Feasibility of ICG-FA for intraoperative assessment of intestinal perfusion | 10 minutes intraoperatively (recording)
  c. Comparison of the number of procedures in which it was a priori possible to perform ICG-FA imaging and the number of procedures in which the device was eventually used intraoperatively (applicability);
Feasibility of ICG-FA for intraoperative assessment of intestinal perfusion | 10 minutes intraoperatively (recording)
  d. Interference with intraoperative Near Infrared Spectroscopy (NIRS) brain monitoring (compatibility: brain monitoring not interfered with/possible despite interference/impossible due to interference);
Safety of intraoperative ICG-FA in gastrointestinal surgery for young infants and neonates | 24 hours
  a. Number of complications directly related to use of the device or extension of operative time for ICG-FA imaging, occurring within 24 hours after surgery in the patients involved in this study;
Safety of intraoperative ICG-FA in gastrointestinal surgery for young infants and neonates | 24 hours
  b. Measurement of the prolonged OR time associated with intraoperative ICG-FA in minutes;

SECONDARY OUTCOMES:
Comparison of conventional and ICG-FA mediated assessment | Through study completion, on average within 4 weeks
  a. Comparing whether the perfusion assessment of ICG-FA can provide more certainty on the perfusion status of intestinal sections than conventional visual assessment (by comparing ICG-FA images with normal view images) in order to identify whether ICG-FA, if applied for decision-making, would have confirmed or altered intraoperative decision making.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Hulscher, MD, PhD, Principal Investigator — UMC Groningen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cahill RA, Ris F, Mortensen NJ. Near-infrared laparoscopy for real-time intra-operative arterial and lymphatic perfusion imaging. Colorectal Dis. 2011 Nov;13 Suppl 7:12-7. doi: 10.1111/j.1463-1318.2011.02772.x. PMID 22098511
- [Background] Jafari MD, Wexner SD, Martz JE, McLemore EC, Margolin DA, Sherwinter DA, Lee SW, Senagore AJ, Phelan MJ, Stamos MJ. Perfusion assessment in laparoscopic left-sided/anterior resection (PILLAR II): a multi-institutional study. J Am Coll Surg. 2015 Jan;220(1):82-92.e1. doi: 10.1016/j.jamcollsurg.2014.09.015. Epub 2014 Sep 28. PMID 25451666
- [Background] Ris F, Liot E, Buchs NC, Kraus R, Ismael G, Belfontali V, Douissard J, Cunningham C, Lindsey I, Guy R, Jones O, George B, Morel P, Mortensen NJ, Hompes R, Cahill RA; Near-Infrared Anastomotic Perfusion Assessment Network VOIR. Multicentre phase II trial of near-infrared imaging in elective colorectal surgery. Br J Surg. 2018 Sep;105(10):1359-1367. doi: 10.1002/bjs.10844. Epub 2018 Apr 16. PMID 29663330
- [Background] Liu D, Liang L, Liu L, Zhu Z. Does intraoperative indocyanine green fluorescence angiography decrease the incidence of anastomotic leakage in colorectal surgery? A systematic review and meta-analysis. Int J Colorectal Dis. 2021 Jan;36(1):57-66. doi: 10.1007/s00384-020-03741-5. Epub 2020 Sep 18. PMID 32944782
- [Background] Lin J, Zheng B, Lin S, Chen Z, Chen S. The efficacy of intraoperative ICG fluorescence angiography on anastomotic leak after resection for colorectal cancer: a meta-analysis. Int J Colorectal Dis. 2021 Jan;36(1):27-39. doi: 10.1007/s00384-020-03729-1. Epub 2020 Sep 4. PMID 32886195
- [Background] Mok HT, Ong ZH, Yaow CYL, Ng CH, Buan BJL, Wong NW, Chong CS. Indocyanine green fluorescent imaging on anastomotic leakage in colectomies: a network meta-analysis and systematic review. Int J Colorectal Dis. 2020 Dec;35(12):2365-2369. doi: 10.1007/s00384-020-03723-7. Epub 2020 Aug 26. PMID 32845390
- [Background] van den Bos J, Al-Taher M, Schols RM, van Kuijk S, Bouvy ND, Stassen LPS. Near-Infrared Fluorescence Imaging for Real-Time Intraoperative Guidance in Anastomotic Colorectal Surgery: A Systematic Review of Literature. J Laparoendosc Adv Surg Tech A. 2018 Feb;28(2):157-167. doi: 10.1089/lap.2017.0231. Epub 2017 Nov 6. PMID 29106320
- [Background] Alekseev M, Rybakov E, Shelygin Y, Chernyshov S, Zarodnyuk I. A study investigating the perfusion of colorectal anastomoses using fluorescence angiography: results of the FLAG randomized trial. Colorectal Dis. 2020 Sep;22(9):1147-1153. doi: 10.1111/codi.15037. Epub 2020 Apr 6. PMID 32189424
- [Background] Wales PW, de Silva N, Kim JH, Lecce L, Sandhu A, Moore AM. Neonatal short bowel syndrome: a cohort study. J Pediatr Surg. 2005 May;40(5):755-62. doi: 10.1016/j.jpedsurg.2005.01.037. PMID 15937809
- [Background] Breuking EA, van Varsseveld OC, Harms M, Tytgat SHAJ, Hulscher JBF, Ruiterkamp J. Safety and Feasibility of Indocyanine Green Fluorescence Angiography in Pediatric Gastrointestinal Surgery: A Systematic Review. J Pediatr Surg. 2023 Aug;58(8):1534-1542. doi: 10.1016/j.jpedsurg.2022.10.045. Epub 2022 Oct 24. PMID 36404183
- [Background] Hirayama Y, Iinuma Y, Yokoyama N, Otani T, Masui D, Komatsuzaki N, Higashidate N, Tsuruhisa S, Iida H, Nakaya K, Naito S, Nitta K, Yagi M. Near-infrared fluorescence cholangiography with indocyanine green for biliary atresia. Real-time imaging during the Kasai procedure: a pilot study. Pediatr Surg Int. 2015 Dec;31(12):1177-82. doi: 10.1007/s00383-015-3799-4. Epub 2015 Oct 6. PMID 26439370
- [Background] Rentea RM, Halleran DR, Ahmad H, Sanchez AV, Gasior AC, McCracken K, Hewitt GD, Alexander V, Smith C, Weaver L, Wood RJ, Levitt MA. Preliminary Use of Indocyanine Green Fluorescence Angiography and Value in Predicting the Vascular Supply of Tissues Needed to Perform Cloacal, Anorectal Malformation, and Hirschsprung Reconstructions. Eur J Pediatr Surg. 2020 Dec;30(6):505-511. doi: 10.1055/s-0039-1700548. Epub 2019 Dec 13. PMID 31858494
- [Background] Clements KE, Fisher M, Quaye K, O'Donnell R, Whyte C, Horgan MJ. Surgical site infections in the NICU. J Pediatr Surg. 2016 Sep;51(9):1405-8. doi: 10.1016/j.jpedsurg.2016.04.002. Epub 2016 Apr 11. PMID 27132541
- [Background] Eeftinck Schattenkerk LD, Musters GD, Nijssen DJ, de Jonge WJ, de Vries R, van Heurn LWE, Derikx JPM. The incidence of abdominal surgical site infections after abdominal birth defects surgery in infants: A systematic review with meta-analysis. J Pediatr Surg. 2021 Sep;56(9):1547-1554. doi: 10.1016/j.jpedsurg.2021.01.018. Epub 2021 Jan 17. PMID 33485614
- [Background] Iinuma Y, Hirayama Y, Yokoyama N, Otani T, Nitta K, Hashidate H, Yoshida M, Iida H, Masui D, Manabe S. Intraoperative near-infrared indocyanine green fluorescence angiography (NIR-ICG AG) can predict delayed small bowel stricture after ischemic intestinal injury: report of a case. J Pediatr Surg. 2013 May;48(5):1123-8. doi: 10.1016/j.jpedsurg.2013.03.067. PMID 23701792
- [Background] Kamran A, Zendejas B, Meisner J, Choi SS, Munoz-San Julian C, Ngo P, Manfredi M, Yasuda JL, Smithers CJ, Hamilton TE, Jennings RW. Effect of Posterior Tracheopexy on Risk of Recurrence in Children after Recurrent Tracheo-Esophageal Fistula Repair. J Am Coll Surg. 2021 May;232(5):690-698. doi: 10.1016/j.jamcollsurg.2021.01.011. Epub 2021 Feb 5. PMID 33556502
- [Background] Meira J, Marques ML, Falcao-Reis F, Rebelo Gomes E, Carneiro A. Immediate Reactions to Fluorescein and Indocyanine Green in Retinal Angiography: Review of Literature and Proposal for Patient's Evaluation. Clin Ophthalmol. 2020 Jan 20;14:171-178. doi: 10.2147/OPTH.S234858. eCollection 2020. PMID 32021082
- See also: Verdye Indocyanine Green description (Dutch) — https://db.cbg-meb.nl/bijsluiters/h31052.pdf